CLINICAL TRIAL: NCT05446402
Title: Double Blinded, Split Face Investigation of the Tolerability of Two Facial Cleansing Routines for Mild to Moderate Acne
Brief Title: Investigation of the Tolerability of Two Facial Cleansing Routines for Mild to Moderate Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stephanie Rangel, Principal Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU#00217056
Record Dates: First submitted 2022-06-30; First posted 2022-07-06 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Participants will be using Product 1 regimen on left side of face for 12 weeks and Product 2 regimen on right side of face for 12 weeks.
Masking Description: All sets of products will be provided to Northwestern in identical, unlabeled bottles for the purpose of blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acne Treatment (Experimental)
  Interventions: Combination Product: Geologie Acne Regimen - one side of face; Combination Product: Proactive Acne Regimen - other side of face

INTERVENTIONS:
Combination Product: Geologie Acne Regimen - one side of face — Geologie is an over-the-counter cosmetic acne regimen with three products. The regimen also has three "levels" over the course of three months, in which the nighttime lotion is switched to a stronger formula each month. The Geologie Clear System regimen for acne prone skin includes:
  1. Clarifying Gel Cleanser - SA Formula (2% Salicylic Acid)
  2. Brightening Day Cream - SPF 15 (5% Azelaic Acid, 2% Hyaluronic Acid, 1%Niacinamide)
  3. Repairing Night Cream -
     1. Level 1 (0.05% Retinol, 3% Niacinamide, 2% Hyaluronic Acid)
     2. Level 2 (0.2% Retinol, 3% Niacinamide, 2% Hyaluronic Acid)
     3. Level 3 (0.3% Retinol, 3% Niacinamide, 2% Hyaluronic Acid)
Combination Product: Proactive Acne Regimen - other side of face — ProActiv is an over-the-counter cosmetic regimen with three products. The
  Proactiv Solution 3-Piece System regimen includes:
  1. Renewing Cleanser (Active ingredient: 2.5% Benzoyl Peroxide)
  2. Revitalizing Toner (Glycolic Acid)
  3. Repairing Treatment (Active ingredient: 2.5% Benzoyl Peroxide)

SUMMARY:
The objective of this study is to compare tolerability of two similar commercially available over the counter acne regimens (Geologie and Proactiv) in individuals with mild to moderate acne vulgaris over a 12-week daily treatment course.

DETAILED DESCRIPTION:
Acne vulgaris is a common, chronic inflammatory skin disorder that originates in the pilosebaceous unit. Acne typically begins in adolescence and often continues into adulthood, with about 20% of cases resulting in scars or hyperpigmentation. It's estimated that acne affects about 85% of adolescents. Individuals who experience acne and acne scars tend to also experience a negative impact on their social and mental health, including depression, anxiety, and social withdrawal. Currently, topical solutions and lifestyle changes are the primary treatment for mild to moderate acne.

This study will evaluate and compare the efficacy of two over the counter products in treating individuals with mild to moderate acne: Geologie and ProActive. Both sets of products will be provided to Northwestern in identical, unlabeled bottles for the purpose of blinding.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* No known active skin infection.
* Presence of mild or moderate acne on face (clinical diagnosis or self-report)
* Willingness to give written consent and comply with study procedures.

Exclusion Criteria:

* Active skin infection.
* Inability to understand instructions or procedures involved.
* Known allergy to ingredient(s) in products being used for study.
* Pregnant women, prisoners, and vulnerable populations.
* Has a history of acute or chronic disease that may interfere with or increase the risk of study participation.
* Has any dermatological disorder that may interfere with the accurate evaluation of the subject's facial appearance, based on the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-06-15 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in IGA Score between Geologie and ProActiv daily treatment | 12 weeks
  Investigator Global Assessment (IGA) will be collected on a scale of 0-4 with 0 being clear and 4 being severe.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Rangel, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No